CLINICAL TRIAL: NCT04143828
Title: MoMiFer-Study: Evaluation of a Mobile Mindfulness Program (mMP) in Individuals/Couples Experiencing Fertility Problems
Brief Title: A Mobile Mindfulness Programme for Individuals/Couples Experiencing Fertility Problems
Acronym: MoMiFer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Katleen Van der Gucht, PhD, Senior Investigator at Leuven Mindfulness Centre - KU Leuven, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S62323
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Infertility
Keywords: Infertility; Mobile Health; Mindfulness
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two conditions: The intervention group receives a mobile mindfulness programme (mMP). The participants in the control group are wait-listed. They will receive access to the mobile mindfulness programme after three months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Mindfulness Programme (Experimental): The mobile mindfulness program is delivered via a mobile application.
  Interventions: Behavioral: mobile mindfulness programme
- Wait-list control condition (No Intervention): When assigned to the control condition, participants will be wait-listed for 3 months during the study. After the final assessment participants will receive access to the mobile mindfulness program.

INTERVENTIONS:
Behavioral: mobile mindfulness programme — The mobile mindfulness programme adheres to a standardized protocol developed from the MBSR curriculum (Kabat-Zinn, 1990). The program consists of six modules. Each module consists of a short movie (talking head) explaining the content and two audiofiles to guide experiential mindfulness meditation exercises. Participants can follow the different modules based on their own time-schedule.
  Key objectives are: (1) to increase awareness of one's present moment experience; (2) to teach an attitude of openness and acceptance (non-judging) toward one's experience.
  Arms: Mobile Mindfulness Programme

SUMMARY:
Infertility and its treatment result in a considerate emotional burden and a recent guideline of the European Society of Human Reproduction (ESHRE) highlight the importance to support couples facing fertility problems. Mindfulness-based programs (MBPs) have been proven effective in improving well-being and combatting mood disturbances in a wide range of conditions in both treatment and prevention. The overall aim of this project is to evaluate the impact of a mobile mindfulness programme (mMP) on quality of life and emotional well-being in individuals/couples experiencing fertility problems. The present study is a two-group randomized controlled trial with assessments at baseline, at 1,5 months and at 3 months. Sixty couples experiencing fertility problems will be enrolled. They will be assigned to either an intervention group (immediate access to the mMP) or a control group (waitlist condition). The mobile MBP is developed by a team of experienced mindfulness trainers, clinical psychologists, and a psychiatrist and adheres to a standardized protocol. The primary outcomes will be quality of life and emotional distress. Secondary outcomes will be repetitive negative thinking, self-compassion and mindfulness skills. Additionally, the feasibility of the mMP will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals/couples experiencing fertility problems (using the criteria for the definition of 'infertility', as in: the failure to achieve a clinical pregnancy after 12 months or more of regular unprotected sexual intercourse) (Zegers-Hochschild et al., 2017)
* Both partners possess a smartphone
* Both partners understand and speak Dutch
* Written informed consent after been informed on all aspects of the study

Exclusion Criteria:

Not applicable

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-24 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Fertility related quality of life | Data collected at baseline (before randomisation), after 1.5 and 3 months
  Change in scores on the Fertility Quality of Life Questionnaire (FertiQol) - 24 items; scoring: 0-100 (the higher the better the quality of life)
emotional distress | Data collected at baseline (before randomisation), after 1.5 and 3 months
  Change in scores on experienced stress, anxiety and depression as measured by Experience Sampling Method (record emotions several times a day during 4 consecutive days); scoring with a sliding bar: 0-100 (the lower the less emotional distress)

SECONDARY OUTCOMES:
repetitive negative thoughts | Data collected at baseline (before randomisation), after 1.5 and 3 months
  Change in scores on the Perseverative Thinking Questionnaire (PTQ) - 15 items; scoring: 0-60 (the higher, the more repetitive negative thinking)
mindfulness skills | Data collected at baseline (before randomisation), after 1.5 and 3 months
  Change in scores on experienced mindfulness skills as measured by Experience Sampling Method (several times a day during 4 consecutive days); scoring with a sliding bar: 0-100 (the higher the better the mindfulness skills)
self-compassion | Data collected at baseline (before randomisation), after 1.5 and 3 months
  Change in scores on the Self Compassion Scale (SCS-NL-R) - 12 items; scoring: 12-60 (the higher the more self-compassion)
Emotional distress | Data collected at baseline (before randomisation), after 1,5 and 3 months
  Change in scores on the Depression, Anxiety and Stress Scale (DASS-21); scoring: 0-126 (the higher the more emotional distress)
Mindfulness skills | Data collected at baseline (before randomisation), after 1,5 and 3 months
  Change in scores on the Comprehensive Inventory of Mindfulness Experiences (CHIME-SF) - 24 items; scoring: 24-144 (the higher the better the mindfulness skills)
subjective quality of the mobile Mindfulness Programme (mMP) | after 3 months in the intervention group
  a shortened version of the subjective quality subscale of the Mobile App Rating Scale (MARS); scoring: 0-8 (the higher, the better the quality of the mMP)
use of the mobile Mindfulness Programme (mMP) | After 1.5 and 3 months in the intervention group
  evaluating the use of the mMP (frequency) in combination with a question on their motivation of (not) using mMP

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Lie Fong, MD. PhD., Principal Investigator — KU Leuven, UZ Leuven; Filip Raes, PhD, Principal Investigator — Leuven Mindfulness Centre - KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
For all the data generated during the course of this project, the investigators will follow the prevailing standards and guidelines in documenting and depositing data sets.
  The investogators will disseminate results from this research through presentations at public lectures, scientific institutions and meetings, and/or publication in major journals. Regarding data sharing, ICMJE recommendations will be followed.
  Individual deidentified participant data will be shared. In particular, individual participant data that underlie the results reported in our articles, after deindentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will become available from 9-36 months after the publication of the RCT-results by the research team.
Access Criteria: Data will only be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Data will be shared to achieve aims in the approved proposal and for individual participant meta-analysis. Proposals should be directed to Katleen.vandergucht@kuleuven.be . To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Boedt T, Willaert N, Lie Fong S, Dancet E, Spiessens C, Raes F, Matthys C, Van der Gucht K. Evaluation of a stand-alone mobile mindfulness app in people experiencing infertility: the protocol for an exploratory randomised controlled trial (MoMiFer-RCT). BMJ Open. 2022 Feb 2;12(2):e050088. doi: 10.1136/bmjopen-2021-050088. PMID 35110309